CLINICAL TRIAL: NCT05462730
Title: Pulse Glucocorticoid Therapy in Patients With ST-Segment Elevation Myocardial Infarction
Acronym: PULSE-MI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thomas Engstrom (Other)
Responsible Party: Sponsor-Investigator, Thomas Engstrom, Professor, MD, Ph.D., DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PULSE-MI; 2022-500762-10-00 (Other: EU-CT number)
Record Dates: First submitted 2022-07-07; First posted 2022-07-18 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: ST Elevation Myocardial Infarction; Inflammatory Response; Myocardial Reperfusion Injury; Myocardial Injury
Keywords: Primary PCI; Inflammation; Reperfusion Injury; Methylprednisolone; Solu-Medrol; Cardioprotection
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Reperfusion Injury; Inflammation; Reperfusion Injury | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, 1:1 randomized, multicenter, double-blind, placebo-controlled clinical trial. A minimum of 378 patients with STEMI will be randomized 1:1 to an infusion of 250 mg (4 mL) methylprednisolone in the pre-hospital setting prior to primary PCI. The methylprednisolone will be given as a bolus infusion of 1 x 250 mg (1 x 4 mL) over a period of 5 minutes. Patients allocated to placebo will receive 4 mL of isotonic saline (NaCl 0.9%).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methylprednisolone (Active Comparator): A five minutes bolus infusion of 250 mg (4 mL) methylprednisolone to inhibit inflammatory damage following ST-segment elevation myocardial infarction. The infusion of methylprednisolone will be given in the pre-hospital setting prior to primary PCI.
  Interventions: Drug: Methylprednisolone
- Isotonic saline (Placebo Comparator): A bolus infusion of 4 mL isotonic saline (NaCl 0.9%).
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Methylprednisolone — A dosis of 250 mg methylprednisolone is suspended in isotonic saline to a total volume of 4 mL prior to infusion.
  Other Names: Solu-Medrol
  Arms: Methylprednisolone
Drug: Isotonic saline — A bolus infusion of 4 mL isotonic saline (NaCl 0.9%).
  Other Names: Isotonic NaCl, Placebo
  Arms: Isotonic saline

SUMMARY:
The overall primary objective of the PULSE-MI trial is to test the hypothesis that administration of single-dose glucocorticoid pulse therapy in the pre-hospital setting reduces final infarct size in patients with ST-segment elevation myocardial infarction (STEMI) treated with primary percutaneous coronary intervention (PCI)

DETAILED DESCRIPTION:
BACKGROUND Myocardial reperfusion with the use of primary percutaneous coronary intervention (PCI) including stent implantation is the most efficacious treatment for patients with (STEMI) and improves prognosis significantly. Due to continuous improvements in the treatment, the mortality for patients with STEMI has decreased dramatically, but despite these improvements, the mortality rate seems to have reached a plateau at around 10% within 1 year. In addition, 10% develop clinical heart failure with a per se 50% mortality rate within 5 years. Moreover, congestive heart failure is associated with a highly impaired quality of life due to fatigue dyspnea and reduced exercise capacity. Thus, there is a need for further improvement in the treatment to drive the event rates further down. One such key target is reducing the damage to the heart muscle (infarct size) to preserve the heart function and prevent mortality and heart failure. One major driver of infarct size is reperfusion injury which may account for up to 50% of the damaged myocardium. Reperfusion injury occurs within the first minutes to hours after the restoration of the blood flow in the occluded artery and reperfusion therapy can therefore be considered a "double-edged sword", since the ischemic injury may additionally be worsened by reperfusion injury. However, the phenomenon of reperfusion injury is not completely understood, and no preventive treatments exist. Multiple pathophysiological factors may contribute to reperfusion injury of which inflammation has been described as a key factor.

Inflammation is induced immediately after the onset of acute myocardial ischemia and is subsequently exacerbated following reperfusion. Hence, inflammation per se may drive excessive cardiomyocyte death resulting in decreased contractility and increased infarct size post-STEMI. Moreover, in the course following STEMI and subsequently reperfusion, the myocardium starts healing and scarring resulting in remodelling of the ventricle potentially causing either compensatory hypertrophy or thinning of the myocardium, which may lead to reduced left ventricle ejection fraction (LVEF) and heart failure. Of note, inflammation plays a critical role in ventricular remodeling post-AMI, thus inflammation in relation to reperfusion injury may extend myocardial damage following STEMI.

Glucocorticoids are crucial in the regulation of the systemic inflammatory response and may therefore be beneficial in limiting myocardial injury following STEMI. Glucocorticoids mediate two different mechanisms: the genomic effect mediated by glucocorticoid receptor occupation, gene transcription, and translation within the cell which is induced within hours, and the non-genomic effect, which is induced rapidly (<15 minutes) after administration via plasma membrane-bound receptors and independent of cytosolic receptor occupation and genomic regulation. Some of the proposed nongenomic effects of glucocorticoids on the cardiovascular system included decreased vascular inflammation and reduced infarct size, cardio protection through membrane stabilisation, and increasing contractility of the vascular smooth muscle cells. Of note, high single-dose glucocorticoid (methylprednisolone) (>250 mg), known as pulse therapy has been proven lifesaving in serval acute conditions including acute rheumatic diseases, exacerbations in lung diseases, imminent cerebral incarceration, and lately COVID-related pulmonary incapacity. The beneficial acute effects of pulse glucocorticoid therapy in these conditions are thought to be mediated by the nongenomic effects of glucocorticoids via plasma membrane-bound receptors, and the estimated complete glucocorticoid receptor occupation is reached at approximately 100 mg methylprednisolone, reaching maximum activation around 250 mg. Moreover, long-term treatment with glucocorticoids is associated with a series of side effects, whereas short-term treatment only has a few side effects. Considering this knowledge of the dual effects of glucocorticoids, safety, and advances in reperfusion strategies, glucocorticoids may now add additional beneficial role in limiting infarct size and improving prognosis in patients with STEMI. Systemic intravenous short-term treatment with glucocorticoids could therefore add an important, beneficial, and safe therapeutic role in limiting the degree of myocardial injury and thereby improving prognosis in patients with STEMI.

In summary, STEMI remains one of the leading causes of mortality globally despite significant advances in reperfusion therapies with timely primary PCI, one in five patients develop heart failure or died within one year following STEMI. The main driver for mortality and heart failure following STEMI is infarct size which is related to ischemia- and reperfusion-induced inflammatory response. Thus, inflammation is an important factor in acute myocardial ischemia and reperfusion injury, which is why inflammation per se is a feasible and desirable target for improving prognosis in these patients. To reduce the degree of inflammation effectively and adequately, intervention is to be made as soon as possible as close to initiation of ischemia, as recognized from patients' symptom debut, and before revascularization with primary PCI in the prehospital setting since the effect is more pronounced if the treatment is initiated early after the onset of STEMI. In addition to reperfusion induced inflammation, ischemia itself, immediately after occlusion of the artery, induces inflammation. Hence, initiation of the intervention in the ambulance is needed to harvest the potentially beneficial and immediate nongenomic effects and subsequent protective genomic actions of pulse glucocorticoid therapy as soon as possible. Thus, by performing intervention in the pre-hospital setting, the investigators expect that participation in the trial will have the potential to produce a direct clinically relevant benefit for the patient resulting in a measurable health-related improvement alleviating the suffering and potentially improving the health of the patient and the prognosis of the medical condition.

HYPOTHESIS In patients with STEMI undergoing primary PCI, 250 mg methylprednisolone administrated in the pre-hospital setting limits reperfusion injury and reduce final infarct size measured by late gadolinium enhancement (LGE) on cardiac magnetic resonance (CMR) 3 months after STEMI.

SAMPLE SIZE The primary endpoint is final infarct size (% of left ventricle mass) measured by LGE on CMR at 3 months. Based on results of the CMR sub-studies of the DANAMI-3 trial, the mean final infarct size measured by LGE on CMR is 13% with a standard deviation (SD) of 9% in patients with STEMI. To demonstrate a relative reduction in final infarct size of 20% with a two-sided alpha level of 0.05 and a power of 80%, recruitment of 378 patients is needed. A drop-out rate of 40% is expected for the primary endpoint. Therefore, the investigators expect to randomize 530 patients in total. However, patients will be included until 378 patients have completed the CMR at 3 months. The power calculations have been calculated by a biostatistics professor.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years including fertile women (It is not possible to perform a pregnancy test (HCG urine test) in the pre-hospital setting. However, methylprednisolone is not contraindicated in pregnant women).
2. Acute onset of chest pain with < 12 hours duration.
3. STEMI as characterized on electrocardiogram (ECG) by one of the following:

1) at least two contiguous leads with ST-segment elevation ≥2.5 mm in men < 40 years, ≥2 mm in men ≥40 years, or ≥1.5 mm in women in leads V2-V3 and/or ≥1 mm in the other leads, 2) presumed new left bundle branch block with ≥1 mm concordant ST-segment ele-vation in leads with a positive QRS complex, or concordant ST-segment depression ≥1 mm in V1-V3, or discordant ST-segment elevation ≥5 mm in leads with a negative QRS complex, 3) Isolated ST depression ≥0.5 mm in leads V1-V3 and ST-segment elevation (≥0.5 mm) in posterior chest wall leads V7-V9 indicating posterior acute myocardial infarc-tion (AMI), 4) ST-segment depression ≥1 mm in eight or more surface leads, coupled with ST-segment elevation in aVR and/or V1 suggesting left main-, or left main equivalent- coronary obstruction.

Exclusion Criteria:

1. Presentation with cardiac arrest (out of hospital cardiac arrest (OHCA)).
2. Time from symptoms onset to primary PCI > 12 hours.
3. Known allergy to glucocorticoid or known mental illness with maniac or psychotic episodes.
4. Patients with previous acute myocardial infarction (AMI) in the assumed culprit artery.
5. Previous coronary artery bypass graft (CABG).
6. Unable to read and understand Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-10-17 (Estimated)

PRIMARY OUTCOMES:
Final Infarct size | 3 months following STEMI
  % of the left ventricle mass measured by late-gadolinium enhancement (LGE) on cardiac magnetic resonance (CMR)

SECONDARY OUTCOMES:
The extent of MVO | During admission
  Microvascular obstruction (MVO) within the LGE identified on CMR
The extent of haemorrhage | During admission
  The extent of haemorrhage identified on T2*-sequences on CMR
CMR efficacy: MVO | During admission
  Microvascular obstruction as a binary outcome (precence/absence): Hypodense areas within the LGE areas
CMR efficacy: Area at risk | During admission
  Visible edema (hypodense areas) on 3D CINE SAX images
CMR efficacy: Extent of Edema | During admission
  hypodense areas on 3D CINE SAX images
CMR efficacy: MSI | During admission and 3 months following STEMI
  Myocardial salvage index (MSI)=infarct size/area-at-risk. MSI will be measured and calculated at the acute CMR and follow-up CMR
CMR efficacy: LVEF | During admission and 3 months following STEMI
  Evaluated on 3D CINE SAX images at the acute and follow-up CMR.
CMR efficacy: Change in infarct size | During admission and 3 months following STEMI
  Calculated as: Follow-up infarct size/acute infarct size. Measured in %.
CMR efficacy: Changes in LVEF | During admission and 3 months following STEMI
  Changes from baseline LVEF to follow-up LVEF on CMR. Measured in %.
Peak Troponin-T and CKMB | During admission
  Peak Troponin-T and CKMB during admission
All-cause mortality and hospitalization for heart failure | 3 months following STEMI
  All-cause mortality and hospitalization for heart failure at 3 months
Safety: Incidence of adverse events | 7 days following admission
  Safety outcome on adverse events

OTHER OUTCOMES:
Pre-PCI and post-PCI TIMI-flow | During primary PCI
  Pre- and post-PCI thrombosis in myocardial infarction (TIMI) flow
CRP, p-glucose, and BNP | During admission
  C-reactive protein (CRP), p-glucose, pro-brain natriuretic peptide (BNP)
LVEF | During admission and 3 months following STEMI
  LVEF on TEE during admission and 3 months following STEMI
Arrythmia | Immediately after discharge
  Ventricular tachycardia/ventricular fibrillation leading to cardioversion from inclusion to hospital discharge
Killip Class | At admission
  Killip Class at admission
Bolus CFR, IMR, absolute CFR and MRR | During primary PCI
  Bolus CFR, IMR, absolute CFR and MRR measured with a pressure wire following primary PCI
Makers of inflammation | At admission, 24 hours after admission, and 3 months after admission
  High sentitivity C-reactive protein (hsCRP), leukocyte- and differential count, plasma cytokine levels (IL-1b, IL-2, IL-4, IL-5, IL-7, IL-8, IL-10, IL-12, IL-13, IL-17A, G-CSF, GM-CSF, MCP-1, MIP-1beta, INF-g, tumor-necrosis factor alfa (TNF-alfa), and procalcitonin
All-cause mortality and hospitalization for HF | 1 year and 10 years following STEMI
  All-cause mortality and hospitalization for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Jacob T Lønborg, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark; Jasmine M Madsen, MD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Heart Center, Rigshospitalet, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marquard JM, Lonborg J, Obling LER, Beske RP, Zhou Y, Nepper-Christensen L, Vejlstrup N, Bang LE, Hassager C, Folke F, Andersen LB, Christensen HC, Holmvang L, Pedersen F, Ahlehoff O, Jabbari R, Minkkinen M, Sorensen R, Tilsted HH, Engstrom T. Prehospital pulse-dose glucocorticoid on index of microvascular resistance in patients with ST-segment elevation myocardial infarction: a sub-study of the PULSE-MI trial. J Inflamm (Lond). 2025 Mar 18;22(1):12. doi: 10.1186/s12950-025-00440-2. PMID 40102868
- [Derived] Madsen JM, Engstrom T, Obling LER, Zhou Y, Nepper-Christensen L, Beske RP, Vejlstrup NG, Bang LE, Hassager C, Folke F, Kyhl K, Andersen LB, Christensen HC, Rytoft L, Arslani K, Holmvang L, Pedersen F, Ahlehoff O, Jabbari R, Barfod C, Hougaard M, Minkkinen M, Tilsted HH, Sorensen R, Lonborg JT. Prehospital Pulse-Dose Glucocorticoid in ST-Segment Elevation Myocardial Infarction: The PULSE-MI Randomized Clinical Trial. JAMA Cardiol. 2024 Oct 1;9(10):882-891. doi: 10.1001/jamacardio.2024.2298. PMID 39211964